CLINICAL TRIAL: NCT01113554
Title: A Pilot Study to Evaluate the Feasibility of a Breast Cancer Rehabilitation Program in Survivors of Breast Cancer
Brief Title: Breast Cancer Rehabilitation Program in Improving Quality of Life in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012783; NCI-2010-00975; CCCWFU 99309 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): Patients attend exercise therapy sessions over 1 hour 3 times a week for 6 months. Exercise therapy sessions are comprised of a 10 minute warm-up of light stretching and aerobic type exercise (walking, cycling), 30 minutes of endurance type exercise (cycle, walking), and 20 minutes of resistance training exercise.
  Interventions: Other: questionnaire administration; Behavioral: exercise intervention; Procedure: quality-of-life assessment; Other: survey administration; Procedure: management of therapy complications; Procedure: psychosocial assessment and care

INTERVENTIONS:
Other: questionnaire administration
Behavioral: exercise intervention
Procedure: quality-of-life assessment
  Other Names: quality of life assessment
Other: survey administration
Procedure: management of therapy complications
  Other Names: complications of therapy, management of
Procedure: psychosocial assessment and care
  Other Names: psychosocial assessment; psychosocial assessment/care; psychosocial care; psychosocial care/assessment; psychosocial studies; psychosocial support

SUMMARY:
RATIONALE: A breast cancer rehabilitation program and exercise therapy may help improve the quality of life of breast cancer survivors.

PURPOSE: This clinical trial studies a breast cancer rehabilitation program in improving quality of life in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate accrual, retention, adherence, and participation of breast cancer survivors to a breast cancer rehabilitation program.

II. To estimate the variability of weight, six-minute walk, quality of life and other psychosocial and physical measures in women participating in the BCRP.

SECONDARY OBJECTIVES:

I. To assess changes in the anthropometric, psychosocial, and physical outcomes over the six-month period of the BCRP.

II. To document the types and the rates of adverse events associated with the BCRP.

OUTLINE:

Patients attend exercise therapy sessions over 1 hour 3 times a week for 6 months. Exercise therapy sessions are comprised of a 10 minute warm-up of light stretching and aerobic type exercise (walking, cycling), 30 minutes of endurance type exercise (cycle, walking), and 20 minutes of resistance training exercise.

ELIGIBILITY:
Inclusion

* First occurrence of breast cancer
* BMI >= 25
* Recently completed treatment(chemotherapy/radiation) for breast cancer (=< 8 weeks), but can be receiving adjuvant hormonal therapy
* Willing to comply with study visits, as outlined in the protocol
* Lives within 30 miles of study site, or willing to travel to study site if outside a 30-mile radius
* Ability to participate in a moderate exercise program, such as freedom from any orthopedic abnormalities that would prevent participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion

* Unstable angina
* Cardiac conduction disturbances
* Plans to move from the study area
* Dementia that is medically documented or suspected
* Advanced arterial disease causing ischemia of any limb
* Physical immobility
* Homebound for medical reasons
* Dependent on wheelchair for mobility
* Chronic disease which significantly reduces 4-year survival
* Recurrent breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Ability to recruit breast cancer survivors into a six-month breast cancer rehabilitation program | Approximately 24 months
BMI | 6 months
Muscular strength | 6 months
Range of motion | 6 months
Quality of life | 6 months
Proportion of screened women who are eligible for the study and the proportion of eligible women who agree to participate | Approximately 24 months
Proportion of women who complete the study and the average number of weeks of participation | Approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mara Vitolins, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States